CLINICAL TRIAL: NCT05073146
Title: Quality Management of Reablement Service by Professionals in Taiwan: Review and Analysis
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202106002RINB
Record Dates: First submitted 2021-08-25; First posted 2021-10-11 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Long-term Care
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: interview — Starting from the user as an extended starting point, through on-site visits and interviews with relevant personnel, such as personal management, professional service teams, cases, family members, other long-term care service providers (home service assistants), etc., collect relevant information and summarize successful strategies and related elements of long-term professional services (including conditions, demand analysis, service usage, professional team interaction, payment and payment systems, characteristics of case, etc.) of model cases.

SUMMARY:
Since the Ministry of Health and Welfare promoted long-term care 2.0 in 2017, it has actively flipped the concept of care. The long-term care professional service added the spirit of self-care, emphasized the dignity and autonomy of the elderly, and provided professional services (including reablement services) to enhance the individual's ability to live independently. However, the use of professional services may be controversial due to unclear understanding of the purpose and service mode of professional services and lack of preparation, vertical (county and city governments, community integrated service centers (A-level units), long-term care service units, etc.) and horizontal cross-professional cooperation is rare, the effectiveness of professional services is unclear, and issues of service quality management also need attention. Therefore, there is an urgent need to integrate the current implementation content and service personnel qualifications of professional services, improve the knowledge of professional service personnel, strengthen the links between county and city governments, A-level units, and long-term care service units, and improve the quality of professional services.

The purpose of this plan is to set up experts and working groups, revise the professional service manuals, develop long-term professional service operation guidelines, review the long-term professional service payment system, and develop professional service quality management mechanisms to provide reference for policy planning.

Researchers will achieve their goals through the following methods:

1. Establish an interdisciplinary, academic and practical expert working group, professional service manual/operation guide revising group, and hold meetings. Researchers will also review professional service manuals and operational guidelines for the drafts of professional services, and the payment system and the improvement mechanism of service quality, etc.
2. Review domestic and foreign documents: four countries including Norway, the United Kingdom, Australia, and Japan. Researchers will compare the long-term care professional service or reablement service models of various countries, and serve as follow-up experts to revise professional service manuals, operating guidelines, and basis for professional service execution and quality management mode.
3. Achievement analysis of model cases: based on the extended case method of qualitative research, it is expected to solicit high-quality model long-term care professional service units, and in-depth collection of relevant information on the characteristics, process and results of the case homes and service units of successful cases of long-term professional services, conduct ethnographic research and benchmarking, understand the operation of the domestic model, as a follow-up reference for the various tasks of this project .
4. Based on the above-mentioned literature review, model case analysis, expert writing, and multiple meetings, develop a long-term professional service manual/long-term professional service operation guidelines, and propose an amendment draft.
5. Suggestions for the review of the payment system for long-term care professional services: methods include the above-mentioned literature review, establishment of an expert group, case visits, analysis of results of typical cases, and discussions on the draft and different payment methods of various care packages and classification of different payment cases, obtain group consensus through the Delphi method, and conduct pros and cons analysis.
6. Conduct simulation verification for the service payment method draft and different payment case classifications, visit cases (including cases with different disability levels or characteristics), and analyze the verification results and make recommendations for revision.
7. Based on the above literature review, analysis of the results of model cases and discussions at expert meetings, develop professional service quality evaluation and management mechanisms
8. Produce public version of long-term professional service manual/long-term professional service operation guide for lecture notes and educational training media, and handle seven sessions of education training in North, Central, South, and East of Taiwan.

ELIGIBILITY:
Clients

Inclusion Criteria:

* (1) The care management specialist or case manager of the A-level unit (community integrated service center) or the B-level unit (combined service center) judged to be an effective professional service user who has reached the age of 20 (e.g. : Decline in the level of disability, decrease in the number of hours of care required, decrease in the burden of caregivers, etc.) and their family members or main caregivers.
* (2) The cognitive status and language ability of professional service users are acceptable for face-to-face (or video) interviews. If the professional service user is a case where a research team such as a dementia patient determines that the cognitive state cannot be interviewed, it will be replaced by interviewing the long-term professional service experience of the family or the main caregiver.
* (3) Understand the research content and agree to accept the interview.

Exclusion Criteria:

* N/A

Caregivers and professionals

Inclusion Criteria:

* (1) The main caregivers of professional service users who have reached the age of 20, and their cognitive and language skills are acceptable for face-to-face (or video) interviews
* (2) Relevant professional service providers (including but not limited to: case managers, care managers, occupational therapists, physiotherapists, nurses, home care service supervisors, caring service supervisor, home service assistants, etc.)
* (3) Understand the research content and agree to accept the interview.

Exclusion Criteria:

* The cognitive status and language ability of the main caregivers in the families of professional service users are not acceptable for face-to-face interviews.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Model cases (long-term professional service users, hereinafter referred to as professional service users, and their family members or main caregivers) and long-term professional service providers of model cases.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Long-Term Care Case-Mix System Score | 5 months
  Collect and analyze participants' Long-Term Care Case-Mix System Score.
Multi-Dimensional Assessment Instrument | 5 months
  Collect and analyze participants' Multi-Dimensional Assessment Instrument Score.

SECONDARY OUTCOMES:
Extended Case interview feedback (Qualitative Research) | 5 months
  Analyze the number of occurrences of specific words in interview transcript.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Medicine, National Taiwan University, Taipei, Taiwan, Taiwan